CLINICAL TRIAL: NCT01529593
Title: Phase I Study of Temsirolimus in Combination With Metformin in Patients With Advanced Cancers
Brief Title: Temsirolimus in Combination With Metformin in Patients With Advanced Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: 75%<Participants
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0923; NCI-2012-00216 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Metastatic cancer; Tumor response; Dose limiting toxicity; DLT; Maximum tolerated dose; MTD; Temsirolimus; CCI-779; Torisel; Metformin
MeSH Terms: conditions — Neoplasm Metastasis | interventions — temsirolimus; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Temsirolimus + Metformin (Experimental): Starting dose of Temsirolimus 25 mg by vein weekly. Metformin titrated over 3 weeks at 500 mg by mouth daily. Four weeks of treatment constitute 1 cycle. Cycle one (1) however, will be 6 weeks long to allow for metformin titration.
  Interventions: Drug: Temsirolimus; Drug: Metformin

INTERVENTIONS:
Drug: Temsirolimus — Starting dose: 25 mg by vein weekly.
  Expansion cohort: Once MTD is determined, or at maximum tolerated dose level explored (Level 5) if MTD is not reached, additional 14 patients enrolled.
  Other Names: CCI-779; Torisel
Drug: Metformin — Starting dose: 500 mg titrated over first 3 weeks.
  Expansion cohort: Once MTD is determined, or at maximum tolerated dose level explored (Level 5) if MTD is not reached, additional 14 patients enrolled

SUMMARY:
This phase I trial studies the side effects and best dose of temsirolimus and metformin hydrochloride in treating patients with cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment (advanced or metastatic). Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Metformin hydrochloride is a drug used to treat diabetes that may also prevent or slow the growth of cancers. Giving temsirolimus and metformin hydrochloride together may kill more tumor cells.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of temsirolimus and metformin based on when you join this study. Up to 6 dose levels of temsirolimus and metformin will be tested. Up to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of the combination of temsirolimus and metformin is found.

Expansion Groups:

When the highest tolerable dose of the study drug combination is found, there will be one group of up to 40 endometrial carcinoma patients enrolled in a tumor-specific expansion group.

Study Drug Administration:

The first study cycle is 42 days and each cycle after that is 28 days. Before you start taking both drugs in Cycle 1, you will take metformin only for the first 2 weeks. This is called a titration period.

On Days 15, 22, 29 and 36 of Cycle 1, you will receive temsirolimus by vein over 30-60 minutes. For each cycle after that, you will receive temsirolimus by vein over 30-60 minutes on Days 1, 8, 15, and 22.

Before you receive temsirolimus, you will receive Benadryl (diphenhydramine) by vein over 30-60 minutes to help lower the risk of allergic reactions.

You will take metformin by mouth every day at about the same time each day with a meal and cup of water (about 8 ounces). You should take it at home except on the days when you have a study visit. On study visit days, you may take the metformin before you receive the temsirolimus. Depending on your dose, you may take metformin 1-3 times daily. Your study doctor will tell you how to take this drug.

If you are taking metformin before you start this study, the study doctor will let you know how often you will take the metformin and if you will skip the titration period visits described below.

You will be given a letter to take to your home doctor(s) about your study drug administration as part of your care provided outside of MD Anderson.

Study Visits:

At every study visit, you will be asked about your health, any other drugs you are taking, and if you have had any side effects.

Exams and tests will be performed before you receive the study drugs that day. Cycle 1 Day 1 tests and exams may not have to be repeated if done within 7 days.

If you are part of the expansion group, within 7 days before Day 1 of Cycle 1:

* Blood (about 2 teaspoons) will be drawn for pharmacodynamic (PD) testing. PD testing measures how the level of study drug in your body may affect the disease.
* If you are part of the expansion group and have a certain mutation, you will have a biopsy for PD testing. The tumor biopsy will be collected using either a fine needle aspiration or a core biopsy, depending on the location and size of the tumor. To perform a core biopsy, a sample of tissue is removed using a hollow core needle that has a cutting edge. To collect a fine needle aspirate, a small amount of tissue is withdrawn through a needle. If you have questions about your mutation status, the doctor can discuss this with you.

On Day 1 of Cycle 1 (titration period):

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 4 teaspoons) will be drawn for routine tests. You will be asked to not eat anything for 8 hours before your blood draw.
* During Week 1 only, urine will be collected for routine tests.

On Day 8 of Cycle 1 (titration period), blood (about 2 teaspoons) will be drawn for routine tests.

On Day 15 and Day 29 of Cycle 1:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* During Week 1 only, urine will be collected for routine tests.

On Day 22 and Day 36 of Cycle 1, blood (about 2 teaspoons) will be drawn for routine tests.

If you are part of the expansion group, on Day 37 of Cycle 1:

* Blood (about 2 teaspoons) will be drawn for PD testing.
* If you are part of the expansion group and have a certain mutation, you will have a biopsy for PD testing.

On Day 1 of Cycles 2 and beyond:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 4 teaspoons) and urine will be collected for routine tests. You will be asked to not eat anything for 8 hours before your blood draw.

On Day 15 of Cycles 2 and beyond, blood (about 2 teaspoons) will be drawn for routine tests.

About every 8 weeks, you will have an x-ray, CT scan, MRI scan, and/or PET/CT scan to check the status of the disease. If the study doctor thinks it is needed, they will be performed more often.

After about 6 months (about 6 cycles) of taking the study drugs, you will have the CT scan or MRI scan every 2-4 cycles if your study doctor thinks it is needed.

Length of Study Participation:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over when you have completed the end-of-study visit.

End-of-Study Visit:

Within 30 days after your last dose of study drugs, you will return to the clinic. The following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) and urine will be collected for routine tests.

If you are part of the expansion group:

* Blood (about 2 teaspoons) will be drawn for PD testing if the disease gets worse.
* If you are part of the expansion group and have a certain mutation, you will have a biopsy for PD testing if the disease gets worse.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced or metastatic cancer that is refractory to standard therapies, who have relapsed after standard therapy, or whose cancers have no standard therapy that induces a complete response (CR) rate of at least 10% or improves survival by at least three months
* Patients must have evaluable or measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Patients must be >= 4 weeks beyond treatment of any chemotherapy, other investigational therapy, hormonal, biological, targeted agents or radiotherapy, and must have recovered to =< grade 1 or previous baseline for each toxicity; exception: patients may have received palliative low dose radiotherapy to the limbs 1-4 weeks before this therapy provided pelvis, sternum, scapulae, vertebrae, or skull were not included in the radiotherapy field; patients who have received non-chemotherapeutic biological agents will need to wait at least 5 half-lives or 4 weeks (wks), whichever is shorter, from the last day of treatment; continuation of hormone replacement therapy is permitted; stable regimens of hormonal therapy i.e. for prostate cancer (e.g. leuprolide, a gonadotropin-releasing hormone [GnRH] agonist), ovarian, or breast cancer are not exclusionary
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Absolute neutrophil count >= 1000/mL
* Platelets >= 75,000/mL
* Creatinine < 1.5 mg/dl in males and < 1.4 in females
* T. Bilirubin </= 1.5 X ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and/or alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2 X ULN (=< 5 X ULN for patients with liver and/or bone metastases)
* Women of child-bearing potential MUST have a negative serum or urine pregnancy test unless prior hysterectomy or menopause (defined as 12 consecutive months without menstrual activity); patients should not become pregnant or breastfeed while on this study; sexually active patients must agree to use contraception prior to study entry, for the duration of study participation, and for 30 days after the last dose
* Ability to understand and willingness to sign a written informed consent document
* Patients in the tumor-specific endometrial carcinoma expansion cohort that have known mutation must be willing to provide consent for biopsies

Exclusion Criteria:

* Patients who are pregnant or breastfeeding
* Uncontrolled intercurrent illness including, but not limited to, active infection requiring hospitalization
* History of hypersensitivity to temsirolimus or metformin
* History of cerebral vascular accident (CVA), myocardial infarction or unstable angina within the previous six months before starting therapy
* New York Heart Association class III or greater congestive heart failure
* Patients with major surgery within 30 days prior to entering the study
* Patients unable to swallow oral medications or with pre-existing gastrointestinal disorders that might interfere with proper absorption of oral drugs
* Patients on drugs that are strong cytochrome P450, family 3, subfamily A, polypeptide 4 (P450 CYP3A4) modifiers; these drugs should be stopped 5 half-lives prior to starting investigational agents with temsirolimus; the strong inducing or inhibiting agents should not restart until 1 week after the end of the study treatment; NOTE: we will allow replacement of steroids (with either prednisone or hydrocortisone) in patients with adrenalectomy
* Patients with a history of any grade of persistent or chronic nausea or vomiting within the last 4 weeks related to prior therapy or disease process

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-03-26 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Temsirolimus and Metformin | 10 weeks
  MTD defined as highest dose studied in which incidence of dose limiting toxicity (DLT) less than 33%. DLTs defined as adverse events (AEs) related to study agents which occur during first cycle of treatment. Toxicity must have possible, probable or definite attribution to study drugs.

SECONDARY OUTCOMES:
Clinical Tumor Response | 10 weeks
  Clinical efficacy measured by objective tumor response per RECIST (Response Evaluation Criteria In Solid Tumors) criteria. Clinical response defined as Complete Response (CR) or Partial Response (PR) or at least 4 months Stable Disease (SD).

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Ahmed J, Stephen B, Khawaja MR, Yang Y, Salih I, Barrientos-Toro E, Raso MG, Karp DD, Piha-Paul SA, Sood AK, Ng CS, Johnson A, Soliman PT, Meric-Bernstam F, Lu KH, Naing A. A phase I study of temsirolimus in combination with metformin in patients with advanced or recurrent endometrial cancer. Gynecol Oncol. 2025 Feb;193:73-80. doi: 10.1016/j.ygyno.2024.12.019. Epub 2025 Jan 8. PMID 39787747
- [Derived] Liu X, Lorusso P, Mita M, Piha-Paul S, Hong DS, Fu S, McQuinn L, Asatiani E, Doyle LA, Chen HX, Hess KR, Kurzrock R, Naing A. Incidence of mucositis in patients treated with temsirolimus-based regimens and correlation to treatment response. Oncologist. 2014 Apr;19(4):426-8. doi: 10.1634/theoncologist.2013-0231. Epub 2014 Mar 25. PMID 24668327
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org